CLINICAL TRIAL: NCT02560337
Title: Cabazitaxel in Patients With Recurrent Ovarian Cancer After Failure of Standard Therapy - A Phase II Trial
Brief Title: Cabazitaxel in Patients With Recurrent Ovarian Cancer After Failure of Standard Therapy.
Acronym: CaTo-ROC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vejle Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CaTo-ROC
Record Dates: First submitted 2015-09-23; First posted 2015-09-25 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Ovarian Cancer
Keywords: Ovarian cancer; Relapse; Recurrence; Chemotherapy resistance
MeSH Terms: conditions — Ovarian Neoplasms; Recurrence | interventions — cabazitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cabazitaxel (Experimental): 25 mg/m2 administered as a one hour intravenous infusion on day 1 of a 3-week cycle.
  Treatment continues until progression or unacceptable toxicity.
  Interventions: Drug: Cabazitaxel

INTERVENTIONS:
Drug: Cabazitaxel
  Other Names: Jevtana

SUMMARY:
Many ovarian cancer patients have been offered different standard cytostatics and gradually develop chemo-resistance. However, a considerable fraction of these patients are still in good general health and have a strong wish for further treatment.

Cabazitaxel (Jevtana®) is a new taxane with effect in breast and prostatic cancer. In both tumors it has shown effect in patients refractory to docetaxel. Therefore, it could be anticipated that cabazitaxel may also have an effect in chemo-resistant ovarian cancer.

The aim of the study is to investigate whether cabazitaxel could be a reasonable treatment option in patients with chemo-resistant and refractory ovarian cancer with regard to effect and toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed epithelial, primary fallopian or primary peritoneal cancer.
* Platinum resistant ovarian cancer with at least two previous cytostatic regimens or platinum-refractory disease defined as progression while receiving the last line of platinum based therapy or within 4 weeks of last platinum dose
* Progression on previous treatment.
* Measurable disease by RECIST 1.1 or evaluable by GCIG CA-125 criteria
* Age ≥ 18 years.
* Performance status 0-2.
* Adequate bone marrow function, liver function, and renal function (within 7 days prior to inclusion):

  * Neutrophils (ANC) ≥ 1.5 * 10^9/l
  * Platelet count ≥ 100 * 10^9/l
  * Hemoglobin ≥ 9.0 g/dL or ≥ 5.6 mmol/l
  * Serum bilirubin ≤ 1.0 * ULN
  * Serum transaminase ≤ 2.5 * ULN
  * Serum creatinine ≤ 1.5 ULN (at creatinine above 1.5 x ULN measured GFR must be at least 50 ml / min)
* Remaining life expectancy of at least 3 months
* Written informed consent

Exclusion Criteria:

* History of severe hypersensitivity reaction (≥grade 3) to taxol.
* History of severe hypersensitivity reaction (≥grade 3) to polysorbate 80 containing drugs.
* Allergy to the active substance or any of the auxiliary agents.
* Concurrent or planned treatment with strong inhibitors or strong inducers of cytochrome P450 3A4/5 (a 2-week wash-out period is necessary for patients who are already on these treatments)
* Neuropathy grade ≥ 2.
* Pregnant or breast-feeding patients. For fertile women a negative pregnancy test at screening is mandatory.
* Fertile patients not willing to use effective methods of contraception during treatment and for 6 months after the end of treatment.
* Other malignant diseases within 5 years prior to inclusion in the study, except basal cell or squamous cell carcinoma of the skin and cervical carcinoma-in-situ.
* Other experimental therapy or participation in another clinical trial within 28 days prior to treatment initiation.
* History of any chronic medical or psychiatric condition or laboratory abnormality that is not medically controlled or in the opinion of the investigator may increase the risks associated with study drug administration. (e.g. diabetes, cardiac diseases, hypertension, renal, thyroid or liver disease).
* Vaccination with yellow fever vaccine or any live attenuated vaccine during the treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-12-05 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Number of patients alive and without progression after three months of treatment | 3 months after start of treatment

SECONDARY OUTCOMES:
Response rate | Every 9 weeks from date of enrollment until the date of first documented progression or date of death of any cause, whichever came first. Assessed up to 24 months
Progression free survival | Every 9 weeks from date of enrollment until the date of first documented progression or date of death of any cause, whichever came first. Assessed up to 24 months
Overall survival | Every three months up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Karina D Steffensen, Study Chair — Vejle Hospital, Department of Oncology
Locations (1):
- Vejle Hospital, Department of Oncology, Vejle, Denmark